CLINICAL TRIAL: NCT01030029
Title: Auricular Acupuncture in Postoperative Pain: a Randomized Controlled Trail
Brief Title: Auricular Acupuncture in Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Department of Anesthesiology, General Intensive Care Medicine and Pain Control (Unknown)
Responsible Party: Andrea Holzer, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08/2009; 262/2005 (Other: ethical commitee)
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2006-01

CONDITIONS: Acupuncture
Keywords: auricular acupuncture; postoperative pain; opioid consumption; laparoscopic surgery; ACUPUNCTURE THERAPY (IM) + EAR, EXTERNAL (IM)
MeSH Terms: conditions — Pain, Postoperative | interventions — Electric Stimulation; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- electrical auricular acupuncture (Active Comparator): Patients in the acupuncture group received titan disposable needles (27-gauge, 3 mm length; Biegler GmbH, Mauerbach, Austria), which were inserted in the dominant ear at the following acupuncture points: shen men, thalamus and one segmental organ-specific point. Acupuncture points were identified by measuring skin resistance, using an electrical conductance meter (multipoint selection pen™, Biegler GmbH, Mauerbach, Austria). The needles were connected to the P-Stim™ device and received continuous low frequency electro acupuncture using P-Stim™ (constant current: 1 Hz biphasic, 2 mA) for 72 hours postoperatively. Acupuncture was performed by a specialist with 15 years experience in this technique.
  Interventions: Device: electrical auricular acupuncture
- pstim device without acupuncture (Placebo Comparator): Patients in the control group received electrodes without needles and the P-Stim™ devices were applied without electrical stimulation.
  Interventions: Device: P-Stim™ devices were applied without electrical stimulation and acupuncture.

INTERVENTIONS:
Device: electrical auricular acupuncture — Patients in the acupuncture group received titan disposable needles (27-gauge, 3 mm length; Biegler GmbH, Mauerbach, Austria), which were inserted in the dominant ear at the following acupuncture points: shen men, thalamus and one segmental organ-specific point [2]. Acupuncture points were identified by measuring skin resistance, using an electrical conductance meter (multipoint selection pen™, Biegler GmbH, Mauerbach, Austria). The needles were connected to the P-Stim™ device and received continuous low frequency electro acupuncture using P-Stim™ (constant current: 1 Hz biphasic, 2 mA) for 72 hours postoperatively. Acupuncture was performed by a specialist with 15 years experience in this technique.
  Other Names: P-Stim® The stimulator consists of a microcontroller and a bit-coded ST62T60BM6 interface, which produce defined waves of electrical stimuli
  Arms: electrical auricular acupuncture
Device: P-Stim™ devices were applied without electrical stimulation and acupuncture. — Patients in the control group received electrodes without needles and the P-Stim™ devices were applied without electrical stimulation.
  Arms: pstim device without acupuncture

SUMMARY:
The effect of acupuncture for postoperative pain control remains controversial. We therefore studied the effects of electrical auricular acupuncture (AA) on postoperative opioid consumption in a randomized, patient-blinded clinical trial.

40 female patients undergoing laparoscopy were included. Anaesthetized patients were randomly assigned to receive AA (shen men, thalamus and one segmental organ-specific point) or electrodes and electrical stimulation for 72 hours. Postoperatively patients received 1 g paracetamol every 6 hours and additional piritramide on demand. A blinded observer obtained the doses of piritramide and the visual analogue pain scores (VAS) at 0, 2, 24, 48, and 72 hours.

It was the aim of our study to find out, whether auricular acupuncture reduces postoperative pain.

DETAILED DESCRIPTION:
Postoperative pain treatment is a major issue in management of surgical patients. Goal of the treatment is a maximal effect with minimal side effects. There are various treatment options, including conventional pharmacological and complementary approaches. Acupuncture is a system with an empirical basis, which has been used in the treatment for centuries. The mechanisms can be partly explained in terms of endogenous pain inhibitory systems. Its use for pain relief has been supported by clinical trials and this has facilitated its use in pain clinics in most countries. Needle acupuncture and other forms of sensory stimulation produce similar physiological changes in humans and mammals, e.g. rhythmic discharges in nerve fibres, and the release of endogenous opioids. Besides acupuncture points located on "meridians" all over the body acupuncture points are also described on the ear. The stimulation of acupuncture points can be achieved by pressure, a mechanical action of needling, or electrical point stimulation. In chronic pain treatment acupuncture has been found to be more effective than other non-pharmacological therapies. Furthermore, continuous electrical stimulation of auricular acupuncture points improves the treatment of chronic cervical pain patients. Finally, acupuncture represents not only a therapeutically beneficial, but also a cost-effective treatment option. Auricular acupuncture is also known to be effective in treatment of acute postoperative pain.

The aim of our study is to investigate in a randomized, prospective, double - blind, and controlled design whether continuous electrical stimulation of auricular acupuncture points results in reduction of postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* female ASA physical status I-III patients undergoing elective gynaecological laparoscopy

  * (surgery in cases of infertility, ovarian cyst removal, adhesiolysis, adnexal surgery,endometriosis, or hysterectomy),
* aged from 18-60 years.

Exclusion Criteria:

* patients with a history of drug abuse,
* regular use of sedatives,
* chronic analgesic medication,
* neurological or psychiatric diseases,
* adverse reaction to sevoflurane or paracetamol,
* ASA physical status > III,
* pacemaker, or a history of acupuncture treatment.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
mean postoperative pain (VAS score) | 0,2,24,48,72 hours

SECONDARY OUTCOMES:
consumption of piritramide postoperatively | 0,2,24,48,72 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Holzer, MD, Principal Investigator — Medical University Vienna, Department of Anesthesiology and General Intensive Care Medicine
Locations (1):
- Medical University Vienna, Vienna, Austria